CLINICAL TRIAL: NCT04731207
Title: Physiologic Changes of Posterior Ocular Segment During the Menstrual Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suthasinee Sinawat, Associate Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HE631585
Record Dates: First submitted 2021-01-23; First posted 2021-01-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Retinal Vascular
Keywords: retinal vascular density; choroidal thickness; optic nerve head; optical coherence tomography; optical coherence tomography angiography; menstrual cycle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy pregnant women (Other): All participants will be investigated by Optovue® in follicular phase, ovulatory phase, luteal phase of menstrual cycle. The investigation will be done between 12 PM and 1 PM at each phase. Urine pregnancy testing was done at first and last visits. LH ovulation test was performed by the participants own. if the ovulation was detected by urine strip test, the participant have to underwent the Optovue® within 48 hours.
  Interventions: Device: Optovue®

INTERVENTIONS:
Device: Optovue® — Optical coherence tomography and optical coherece tomography angiography

SUMMARY:
Changes of luteinizing hormone (LH), estrogen and progesterone during the menstrual cycle influence the ocular physiology in both anterior and posterior segments. From the literature review, there were no significant differentiation in tear physiology, anterior chamber dept, lens thickness and refractive status. Some studies demonstrated then the central corneal thickness was thinner in the follicular phase, but this is non-conclusive. Advance in ophthalmic technologies provide few studies of posterior segment changes during the menstrual cycle, however, there were quite difference in methodology such as detection methods of ovulation.

DETAILED DESCRIPTION:
There were 2 studies of posterior segment changes during the menstrual cycle. Akar et al showed significant decrease of neuroretinal rim area and increase of cupt area in late luteal phase. Ulas et al found that choroidal thickness was significant thicker in mid-luteal phase. However, the study of retinal vascular density by optical coherence tomography angiography (OCTA) during the menstrual cycle has never been published before.

ELIGIBILITY:
Inclusion Criteria:

* Female with age 25-40 yr
* Normal body mass index (18.5-24.9)
* Regular menstrual cycle (28-32 days)
* Written informed consent

Exclusion Criteria:

* Pregnant women
* Lactating women
* Having childbirth or miscarriage within 6 months
* Systemic diseases which need taking the regular medication
* History of ocular disease such as glaucoma, retinal vascular diseases and macular disease
* History of hormonal taking such as oral contraceptive pills within 6 months
* History of intraocular laser and intraocular surgery
* Refractive error; spherical equivalent >4 diopters
* Can not taking the images by Optovue® such as spine diseases

Withdrawal criteria

* Pregnancy detection during the study period
* Receiving sex hormone during the study period such as emergency contraceptive pills

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Retinal vascular density | 1 month
  % of retinal vascular density is measured by optical coherence tomography angiography

SECONDARY OUTCOMES:
Choroidal thickness | 1 month
  Choroidal thickness (um) is measured by optical coherence tomography
Retinal nerve fiber layer thickness | 1 month
  Retinal nerve fiber layer thickness (um) is measured by optical coherence tomography
Optic nerve head topography | 1 month
  Disc area and cup area (mm3) are measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, MD, Principal Investigator — KKU Eye Center, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No